CLINICAL TRIAL: NCT00237185
Title: Open, Randomized, Phase II Study of Glivec in Patients With Unresectable or Metastatic Gastrointestinal Stromal Tumors Expressing C-kit Plus 10 Year Extension Study
Brief Title: A Study of the Efficacy and Safety of Imatinib Mesylate in Patients With Unresectable or Metastatic Gastrointestinal Stromal Tumors Expressing C-kit Gene
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571B2222; CSTI571B2222/E1
Record Dates: First submitted 2005-10-09; First posted 2005-10-12 (Estimated); Results first posted 2014-07-15 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Unresectable or Metastatic Malignant Gastrointestinal Stromal Tumor (GIST)
Keywords: GIST; c-kit; imatinib mesylate
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Piebaldism | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- imatinib mesylate 400 mg (Experimental): 400 mg once daily
  Interventions: Drug: Imatinib mesylate
- imatinib mesylate 600 mg (Experimental): 600 mg once daily
  Interventions: Drug: Imatinib mesylate

INTERVENTIONS:
Drug: Imatinib mesylate — Participants were randomized 1:1 to receive imatinib mesylate 400 mg/day or 600 mg/day. Upon unsatisfactory treatment effect on the starting dose of 400 mg/day or 600 mg/day imatinib mesylate, in the opinion of the treating physician, a dose increase up to 600 mg/day or 800 mg/day, was allowed provided that the participant continued to benefit from the treatment and in the absence of safety concerns.
  Other Names: Glivec, Gleevec

SUMMARY:
In the core study, participants with unresectable or metastatic gastrointestinal stromal tumors expressing c-kit were treated with either 400 mg or 600 mg imatinib mesylate for 3 years. The 10 year extension study allowed participants, who successfully completed the core study, to continue study treatment with imatinib mesylate provided they still benefited from treatment and did not demonstrate safety concerns as per the investigator's opinion.

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant women ≥18 years of age with the histopathologically documented diagnosis of malignant GIST that was unresectable and/or metastatic. Confirmation of KIT (CD117) expression via immunohistochemical analysis of tumor sample was also required
* At least one measurable lesion, as defined by Southwestern Oncology Group (SWOG) Solid Tumor Response Criteria, which had not been previously embolized or irradiated
* Performance status ≤3 as defined by the Eastern Cooperative Oncology Group (ECOG) criteria, as well as a life expectancy ≥6 months and adequate end organ function defined as follows: Total bilirubin <1.5 times upper limit of normal (ULN), aspartate aminotransferase (SGOT) and alanine aminotransferase (SGPT) <2.5 x ULN (or <5 x ULN if hepatic metastases were present), creatinine <1.5 x ULN, absolute neutrophil count (ANC) >1.5 x 10^9/L, platelet count >100 x 10^9/L

Exclusion Criteria:

* Patients with fewer than five years of disease-free survival from any other (non-GIST) malignancy except if the other malignancy was not currently clinically significant and did not require active intervention or if the other malignancy was a basal cell skin cancer or a cervical carcinoma in situ
* Patients with known brain metastases
* Evidence of any of the following disorders: Grade III/IV cardiac failure as defined by the New York Heart Association Criteria, severe concomitant disease, acute or known chronic liver disease (i.e. chronic active hepatitis, cirrhosis) or HIV infection
* Chemotherapy or other investigational therapy within four weeks prior to study entry (six weeks for nitrosourea or mitomycin-C) and/or radiotherapy to ≥25% of the bone marrow
* Inability to cooperate
* Major surgery within two weeks or exposure to other investigational agents within 28 days of entry into the study

Other protocol-defined inclusion / exclusion criteria may have applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2000-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Study Chair — Novartis
Locations (5):
- United States (3):
  - Dana Farber Cancer Institute Dept of Sarcoma Oncology, Boston, Massachusetts
  - Oregon Health Sciences University Dept. of Oregon Health Sci., Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Novartis Investigative Site, Geelong, Victoria, Australia
- Novartis Investigative Site, Helsinki, Finland

RESULTS

PARTICIPANT FLOW:
Groups:
- Imatinib Mesylate 400 mg: imatinib mesylate 400 mg once daily
- Imatinib Mesylate 600 mg: imatinib mesylate 600 mg once daily
Period: Core
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Started | 74 | 74
Treated Participants | 73 | 74
Completed | 30 | 37
Not Completed | 44 | 37
Not completed — Adverse Event | 3 | 4
Not completed — Abnormal laboratory value | 0 | 4
Not completed — Abnormal test procedure results | 1 | 0
Not completed — Lack of Efficacy | 30 | 23
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Administrative problems | 0 | 1
Not completed — Death | 4 | 0
Not completed — Determined ineligible post randomization | 1 | 0
Period: Extension
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Started | 24 (A portion of the participants, who completed the core, entered the extension.) | 32 (A portion of the participants, who completed the core, entered the extension.)
Completed | 8 | 13
Not Completed | 16 | 19
Not completed — Adverse Event | 1 | 0
Not completed — Abnormal laboratory value | 0 | 1
Not completed — Lack of Efficacy | 9 | 14
Not completed — Condition no longer required study drug | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Administrative problems | 1 | 0
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Imatinib Mesylate 400 mg: 400 mg
  Imatinib mesylate
- Imatinib Mesylate 600 mg: 600 mg
  Imatinib mesylate
- Total: Total of all reporting groups
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg | Total
Number analyzed (Participants) | 73 | 74 | 147
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (12.9) | 52.2 (11.12) | 54.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 35 | 64
  Male | 44 | 39 | 83

OUTCOME MEASURES:

1. Primary Outcome: Best Tumor Response (Core)
Description: Best tumor response was based on the Southwestern Oncology Group (SWOG) criteria. Objective tumor response assessments were categorized according to the following criteria: complete response (CR), partial response (PR), no change or stable disease (SD), progression of disease (PD), unknown where the progression has not been documented and one or more measurable or evaluable sites have not been assessed (UNK), status after resection for progression (RP), status after resection for safety (RS), status after preventive resection (RPR), progressive after first resection (PDR) and not evaluable. Any tumor assessment after surgical resection for preventative reasons was treated like tumor assessments of UNK for calculation of best response. Tumor assessments with current objective status = RP, RS or PDR were treated like assessments with objective tumor status = PD n the calculation of best response.
Time Frame: Month 36
Population: Treatment population: The treatment population included all randomized participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Number analyzed (Participants) | 73 | 74
participants
  Complete response | 0 | 1
  Partial response | 49 | 49
  Stable disease | 10 | 13
  Progressive disease | 12 | 6
  Not evaluable | 2 | 3
  Unknown | 0 | 2

2. Primary Outcome: Best Tumor Response (Core + Extension)
Description: as for outcome 1
Time Frame: Month 156
Population: Treatment population: the treatment population included all participants who had at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Number analyzed (Participants) | 73 | 74
participants
  Complete response | 1 | 2
  Partial response | 49 | 48
  Stable disease | 10 | 13
  Progressive disease | 11 | 6
  Not evaluable | 2 | 3
  Unknown | 0 | 2

3. Secondary Outcome: Overall Survival (Core)
Description: Overall survival was analyzed as time to event for all participants. Participants who did not die were censored at the last date known alive, which is the last date of any study medication, laboratory sample, tumor assessment, adverse event end date or date of last contact.
Time Frame: Date of first imatinib dose to the date of death during the core period, up to 36 months.
Population: Treatment population: the treatment population included all participants who had at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Number analyzed (Participants) | 73 | 74
months | NA [NA to NA] — The median survival had not been reached. | NA [NA to NA] — The median survival has not been reached.

4. Secondary Outcome: Overall Survival (Core + Extension)
Description: as for outcome 3
Time Frame: Date of first imatinib dose to the date of death during the core and extension periods, up to 156 months.
Population: Treatment population: the treatment population included all participants who had at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Number analyzed (Participants) | 73 | 74
months | 55.9 [34.6 to 85.9] | 57.1 [43.8 to 99.7]

5. Secondary Outcome: Duration of Response (Core)
Description: Duration of response was analyzed as time to event for all participants whose best response was at least a PR. The onset of response was the first tumor assessment that was subsequently confirmed to constitute at least a partial best response. The end of response was the first tumor assessment noting PD.
Time Frame: Date of confirmed best PR or CR to date of confirmed disease progression during the core period, up to 36 months.
Population: Treatment population: the treatment population included all participants who had at least one dose of study medication and whose best response was at least a PR.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Number analyzed (Participants) | 49 | 50
weeks | 113 [83 to NA] — There were not enough events (CRs and PRs) to calculate the upper limit. | 123 [79 to NA] — There were not enough events (CRs and PRs) to calculate the upper limit.

6. Secondary Outcome: Duration of Response (Core + Extension)
Description: as for outcome 5
Time Frame: Date of confirmed best PR or CR to date of confirmed disease progression during the core and extension periods, up to 156 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Number analyzed (Participants) | 49 | 50
months | 27 [22 to 46] | 30 [18 to 56]

7. Secondary Outcome: Progression Free Survival (PFS) (Core + Extension)
Description: Progression free survival was analyzed as a time to event for each participant. If a participant had no event, then the PFS was censored at the last tumor assessment.
Time Frame: Date of first imatinib dose to earliest date of progression, resection due to safety/progression, death due to any cause or discontinuation due to unsatisfactory therapeutic effect during the core and extension periods, up to 156 months.
Population: Treatment population: the treatment population included all participants who had at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Number analyzed (Participants) | 73 | 74
months | 19.3 [16.4 to 28.9] | 25.2 [16.4 to 33.8]

8. Secondary Outcome: Time to Treatment Failure (Core)
Description: Time to treatment failure was analyzed as time to event for all participants. Participants who had neither progressed, died nor discontinued from the trial for any reason other than the condition no longer required therapy were censored for analysis ate the time of their last tumor assessment.
Time Frame: Date of first imatinib dose to date of earliest occurrence of progression, death due to any cause, or discontinuation from the trial for any reason other than the condition no longer required therapy during the core period, up to 36 months.
Population: Treatment population: the treatment population included all participants who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Number analyzed (Participants) | 73 | 74
weeks | 84 [71 to 107] | 84 [71 to 144]

9. Secondary Outcome: Time to Treatment Failure (Core + Extension)
Description: Time to treatment failure was analyzed as time to event for all participants. Participants who had neither progressed, died nor discontinued from the trial for any reason other than the condition no longer required therapy were censored for analysis at the time of their last tumor assessment.
Time Frame: Date of first imatinib dose to date of earliest occurrence of progression, death due to any cause, or discontinuation from the trial for any reason other than the condition no longer required therapy during the core and extension periods, up to 156 month.
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Number analyzed (Participants) | 73 | 74
months | 19 [16 to 25] | 19 [16 to 33]

10. Secondary Outcome: Time to Onset of Response (Core)
Description: Time to response was analyzed as time to event for all participants. Participants who did not meet the definition of confirmed PR/CR were censored at the time of their last progression-free tumor assessment.
Time Frame: Date of first imatinib dose to the date of the first tumor assessment that was later confirmed to be at least a partial response during the core period, up to 36 months.
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Number analyzed (Participants) | 73 | 74
weeks | 13 [12 to 24] | 12 [12 to 22]

11. Secondary Outcome: Time to Onset of Response (Core + Extension)
Description: as for outcome 10
Time Frame: Date of first imatinib dose to the date of the first tumor assessment that was later confirmed to be at least a partial response during the core and extension periods, up to 156 months.
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Number analyzed (Participants) | 73 | 74
months | 3 [3 to 6] | 3 [3 to 3]

12. Secondary Outcome: Time to Progression (Core + Extension)
Description: Time to progression was analyzed as time to event for all participants. Participants who had neither progressed, died nor discontinued from the trial for any reason other than the condition no longer required therapy were censored for analysis at the time of their last tumor assessment.
Time Frame: Date of first imatinib dose to date of progression or death due to disease indication or discontinuation due to unsatisfactory therapeutic effect during the core and extension periods, up to 156 months.
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Number analyzed (Participants) | 73 | 74
months | 19.8 [16.4 to 29.0] | 25.5 [16.5 to 41.5]

ADVERSE EVENTS:
Groups:
- Imatinib Mesylate 400 mg: 400 mg
- Imatinib Mesylate 600 mg: 600 mg
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 600 mg
Serious Adverse Events (participants affected / at risk) | 46/73 | 40/74
Other Adverse Events (participants affected / at risk) | 72/73 | 73/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate 400 mg (N=73) | Imatinib Mesylate 600 mg (N=74)
Anaemia NOS (Blood and lymphatic system disorders) | 2 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 5 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colovesical fistula (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea NOS (Gastrointestinal disorders) | 0 | 2
Diverticular perforation NOS (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 3 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Inflammatory bowel disease NOS (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction NOS (Gastrointestinal disorders) | 2 | 2
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Pancreatitis NOS (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction NOS (Gastrointestinal disorders) | 3 | 2
Vomiting NOS (Gastrointestinal disorders) | 1 | 2
Anasarca (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Disease progression NOS (General disorders) | 1 | 1
Inflammation NOS (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain NOS (General disorders) | 0 | 1
Pain exacerbated (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 2
Rigors (General disorders) | 1 | 0
Cholangitis NOS (Hepatobiliary disorders) | 0 | 1
Cholecystitis NOS (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Abdominal abscess NOS (Infections and infestations) | 1 | 0
Abscess intestinal (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Bronchopneumonia NOS (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Klebsiella infection NOS (Infections and infestations) | 1 | 0
Lung infection NOS (Infections and infestations) | 1 | 0
Orchitis NOS (Infections and infestations) | 1 | 0
Pneumonia NOS (Infections and infestations) | 1 | 1
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Pseudomonas infection NOS (Infections and infestations) | 0 | 1
Sepsis NOS (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Urinary tract infection NOS (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Intestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Postoperative haematoma (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound NOS (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition NOS (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis NOS (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Leukaemia NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anoxic encephalopathy (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Convulsions NOS (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Guillain Barre syndrome (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure NOS (Renal and urinary disorders) | 0 | 2
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Contusion (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash NOS (Skin and subcutaneous tissue disorders) | 1 | 0
Hysterectomy (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
Lung operation NOS (Surgical and medical procedures) | 0 | 1
Operation NOS (Surgical and medical procedures) | 7 | 6
Radiofrequency ablation (Surgical and medical procedures) | 0 | 1
Tracheostomy (Surgical and medical procedures) | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Haemorrhage NOS (Vascular disorders) | 0 | 1
Peripheral vascular disorder NOS (Vascular disorders) | 1 | 0
Petechiae (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib Mesylate 400 mg (N=73) | Imatinib Mesylate 600 mg (N=74)
Anaemia NOS (Blood and lymphatic system disorders) | 12 | 13
Leukopenia NOS (Blood and lymphatic system disorders) | 4 | 5
Neutropenia (Blood and lymphatic system disorders) | 6 | 7
Conjunctival haemorrhage (Eye disorders) | 3 | 6
Conjunctival hyperaemia (Eye disorders) | 2 | 4
Eye irritation (Eye disorders) | 4 | 3
Eyelid oedema (Eye disorders) | 5 | 6
Lacrimation increased (Eye disorders) | 12 | 13
Vision blurred (Eye disorders) | 6 | 2
Abdominal discomfort (Gastrointestinal disorders) | 6 | 9
Abdominal distension (Gastrointestinal disorders) | 7 | 11
Abdominal pain NOS (Gastrointestinal disorders) | 26 | 25
Abdominal pain upper (Gastrointestinal disorders) | 15 | 11
Constipation (Gastrointestinal disorders) | 7 | 7
Diarrhoea NOS (Gastrointestinal disorders) | 43 | 51
Dyspepsia (Gastrointestinal disorders) | 11 | 11
Flatulence (Gastrointestinal disorders) | 22 | 25
Frequent bowel movements (Gastrointestinal disorders) | 2 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 8
Loose stools (Gastrointestinal disorders) | 9 | 7
Nausea (Gastrointestinal disorders) | 45 | 54
Vomiting NOS (Gastrointestinal disorders) | 27 | 25
Asthenia (General disorders) | 4 | 2
Chest pain (General disorders) | 1 | 4
Fatigue (General disorders) | 35 | 39
Influenza like illness (General disorders) | 2 | 4
Lethargy (General disorders) | 4 | 3
Oedema NOS (General disorders) | 7 | 13
Oedema peripheral (General disorders) | 27 | 24
Pain NOS (General disorders) | 3 | 7
Pyrexia (General disorders) | 16 | 11
Rigors (General disorders) | 7 | 5
Gastroenteritis viral NOS (Infections and infestations) | 0 | 4
Influenza (Infections and infestations) | 4 | 3
Nasopharyngitis (Infections and infestations) | 15 | 20
Sinusitis NOS (Infections and infestations) | 4 | 3
Upper respiratory tract infection NOS (Infections and infestations) | 10 | 13
Urinary tract infection NOS (Infections and infestations) | 2 | 8
Liver function test abnormal (Investigations) | 4 | 5
Weight decreased (Investigations) | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 19
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Muscle cramp (Musculoskeletal and connective tissue disorders) | 34 | 43
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 9
Dizziness (Nervous system disorders) | 9 | 7
Dysgeusia (Nervous system disorders) | 2 | 11
Headache (Nervous system disorders) | 22 | 29
Hypoaesthesia (Nervous system disorders) | 2 | 4
Anxiety (Psychiatric disorders) | 8 | 5
Depression (Psychiatric disorders) | 4 | 3
Insomnia (Psychiatric disorders) | 14 | 13
Bronchitis NOS (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 5
Contusion (Skin and subcutaneous tissue disorders) | 4 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 4
Erythema (Skin and subcutaneous tissue disorders) | 1 | 4
Face oedema (Skin and subcutaneous tissue disorders) | 5 | 8
Periorbital oedema (Skin and subcutaneous tissue disorders) | 39 | 39
Photosensitivity reaction NOS (Skin and subcutaneous tissue disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 6
Rash NOS (Skin and subcutaneous tissue disorders) | 24 | 33
Sweating increased (Skin and subcutaneous tissue disorders) | 4 | 2
Flushing (Vascular disorders) | 6 | 5

LIMITATIONS AND CAVEATS:
No safety data was collected in the extension.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.